CLINICAL TRIAL: NCT06770634
Title: Investigation of the Prevalence of Central Sensitization and Associated Factors in Patients With Lipedema
Brief Title: Investigation of Central Sensitization and Associated Factors in Patients With Lipedema
Status: Recruiting | Type: Observational
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Other Study IDs: 2024/14/14/10
Record Dates: First submitted 2025-01-01; First posted 2025-01-13 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Lipedema; Central Sensitisation
Keywords: central sensitization; Lipedema
MeSH Terms: conditions — Lipedema | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- lipedema: patients with lipedema
  Interventions: Other: Pain-Pressure Threshold Measurement With an Algometer; Other: Central Sensitization Inventory; Other: Numeric Rating Scale; Other: Lower Extremity Functional Scale; Other: Short form 12; Other: lower extremity volumetric measurement; Other: lower extremity circumference measurement; Other: Bioelectrical Impedance Analysis; Diagnostic Test: Ultrasound
- Healthy control: Healthy volunteers
  Interventions: Other: Pain-Pressure Threshold Measurement With an Algometer; Other: Central Sensitization Inventory; Other: Lower Extremity Functional Scale; Other: Short form 12; Other: lower extremity circumference measurement; Other: Bioelectrical Impedance Analysis; Diagnostic Test: Ultrasound

INTERVENTIONS:
Other: Pain-Pressure Threshold Measurement With an Algometer — The measurement will be performed 2 times with 3 min intervals for each region and the average of these applications will be recorded. Before the test, a trial test will be applied to the patient. With the pressure algometer, pressure will be applied to the selected points until it causes pain and the test will be terminated for that region when the patient feels pain.
  The measurement includes bilateral thigh, pretibial region and left forearm as remote site and Wagner manual pressure algometer (1 cm2 probe-10 kg/20 lb) will be used. The selected points will be:
  Bilateral thigh: Mid-thigh anterior surface Bilateral pretibial region: Anterior proximal 1/3 of the pretibial area Bilateral forearm volar side center as control point
Other: Central Sensitization Inventory — The central sensitization scale was developed primarily to detect central sensitization findings in patients with chronic pain and consists of two parts, A and B. In part A, 25 somatic and psychosocial symptoms frequently found in patients with central sensitization.
  Other Names: CSI
Other: Numeric Rating Scale — Leg pain, feeling of tension and heaviness on the affected arm will be evaluated separately by numerical scale.
  Groups: lipedema
Other: Lower Extremity Functional Scale — The lower extremity functional scale is a valid patient-rated outcome measure for the measurement of lower extremity function. The scale consist of 4 groups with 20 questions. The questions in these group focus on activities with increasing physical demands like questions from walking between rooms to running on uneven ground. The scoring of this scale varies from 0 (extreme difficulty/unable to perform activity) to 4 (no difficulty). The total score can be obtained by summing the scores of the individual items. The maximum score of 80 indicates no functional limitations and the minimum score of 0 indicates extreme limitations.
  Other Names: LEFS
Other: Short form 12 — The Short form 12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure.The scoring yields two summary measures: the Physical Component Summary (PCS) and the Mental Component Summary (MCS).Utilize the norm-based scoring system to interpret PCS and MCS scores, with a mean of 50 and a standard deviation of 10 in the general population.Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Other: lower extremity volumetric measurement — It is calculated by converting the circumference measurements taken at 4 cm intervals from the ankle to the proximal thigh into lower extremity volume with Excel.
  Groups: lipedema
Other: lower extremity circumference measurement — bilateral tuberosity tibia, 20 cm proximal tuberosity tibia, tuberosity tibia 10 cm distal and ankle level
Other: Bioelectrical Impedance Analysis — With Bioelectrical Impedance Analysis, fat, muscle and water ratio and lean mass are calculated in addition to the patient's body weight.
Diagnostic Test: Ultrasound — Measurement of subcutaneous fat tissue thickness from mid-thigh, pretibial, lateral leg and supramalleolar regions with ultrasound.The average of two measurements taken from the same area will be recorded.According to these measurements; 12-15 mm = mild lipedema or lipohyperplasia, 15-20 mm = moderate lipedema, >20 mm = significant lipedema, >30 mm = severe lipedema.

SUMMARY:
This study aims to investigate the presence of central sensitization and its associated parameters in patients with lipedema. Lipedema is a chronic and hereditary condition that primarily affects the lower extremities in women and is often associated with hormonal changes. Symptoms such as pain, swelling, and tenderness are common in lipedema, and these symptoms may be related to central sensitization. Additionally, the ultrasonographic findings and pain sensitivity in lipedema will be compared with those of healthy individuals. This study seeks to contribute to the diagnosis and treatment process of lipedema.

DETAILED DESCRIPTION:
Lipedema is a chronic and hereditary condition that affects the subcutaneous fat tissue, particularly in the lower extremities of women. Although its prevalence is not clearly known, it is estimated to be common in the general population. It typically begins during periods of weight gain associated with hormonal changes such as puberty, pregnancy, and menopause. It is characterized by persistent swelling in the lower extremities, especially in the upper thighs, which does not improve with elevation, and is painful to touch. Patients often report easy bruising even with minor trauma or touch. The hips and gluteal region are the most commonly affected areas, and the hands and feet are typically spared. On examination, the affected extremities feel soft and doughy due to fat hypertrophy, and there is an increased sensitivity across the area. During follow-up, patients' weight and body mass index (BMI) should be monitored, and the circumferences and volumes of the affected extremities should be measured and recorded.

The diagnosis is usually made clinically after ruling out other differential diagnoses. Among the auxiliary imaging methods, ultrasound (US), computed tomography (CT), and magnetic resonance imaging (MRI) can be used to evaluate the skin and subcutaneous fat tissue. US is frequently preferred in the diagnosis of lipedema as it allows differentiation from lymphedema. Common ultrasonographic findings of lipedema include normal skin thickness, increased thickness of the subcutaneous layer, homogeneous expansion of this layer, and a decrease in echogenicity. A key issue in the diagnosis of lipedema is its confusion with obesity, a prevalent health issue in the general population.

Pain is a significant symptom in patients with lipedema. Studies have shown that pain and increased sensitivity in the swollen extremities of lipedema patients negatively affect their quality of life. Patients frequently complain of nonspecific pain and tenderness, thought to be transmitted by A beta and C fibers, a phenomenon known as allodynia. These complaints are believed to be associated with an increase in pain sensitivity.

Central sensitization is the increased sensitivity of the central nervous system to pain. This condition is associated with exaggerated pain responses to stimuli from specific areas of the body, especially in patients with chronic pain. The pain experienced in lipedema, which worsens even with mild stimuli like touch, raises the possibility of central sensitization. These findings suggest that pain in lipedema is not merely a localized fat tissue issue, but rather a complex process that also affects the nervous system. Therefore, although the presence of central sensitization in lipedema has not been conclusively proven, it is believed that central sensitization may occur in lipedema, considering the role of chronic pain and neurogenic mechanisms. This study aims to investigate the presence of central sensitization and its associated parameters in patients with lipedema. Additionally, the study will examine the differences and similarities in ultrasonographic and pain sensitivity findings between individuals with lipedema and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

1. Lipedema; Diagnosis of lipedema Aged between 18 and 65 years Literate Willing to participate in the study
2. control group; Being completely healthy (no internal/metabolic issues such as diabetes, obesity, or hypothyroidism, and no diagnosis of lipedema) BMI ≤ 30 Aged between 18 and 65 years Literate Willing to participate in the study

Exclusion Criteria:

1. Lipedema group; Under 18 or over 65 years of age Presence of concurrent lymphedema, chronic venous insufficiency, deep vein thrombosis, polyneuropathy, or fibromyalgia Illiterate Not willing to participate in the study
2. Control group; Under 18 or over 65 years of age Presence of concurrent lymphedema, chronic venous insufficiency, deep vein thrombosis, polyneuropathy, fibromyalgia, systemic rheumatic diseases, active cancer, infections, or pregnancy Illiterate Not willing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our study will be conducted as a cross-sectional, single-center study with lipedema-diagnosed patients and healthy volunteers who apply to the Physical Medicine and Rehabilitation outpatient clinic of Sultan 2nd Abdülhamid Han Hospital, Health Sciences University. Participants who meet the inclusion and exclusion criteria will be asked to complete the specified scales. In addition to clinical parameters, ultrasonographic evaluation and pressure pain threshold measurement using an algometer will be performed.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Central Sensitization Inventory | 3 months
  The Central Sensitization Inventory (CSI) is a tool used to assess the heightened sensitivity of the central nervous system. This scale is designed to identify the effects of central sensitization commonly seen in chronic pain conditions by examining an individual's pain perception, sensory changes (such as sensitivity to heat, cold, or pressure), the impact of persistent pain on daily activities, and the emotional effects of pain (such as anxiety, depression, etc.). It plays a crucial role in both clinical practice and research for diagnosing chronic pain syndromes and monitoring treatment responses.
Pressure Pain Threshold | 3 months
  The purpose of this test is to measure the pressure pain threshold, defined as the minimal pressure level that causes pain. The test will be performed twice for each region with a 3-minute interval, and the average of these measurements will be recorded. Before the test, a trial run will be conducted for the patient. Using a pressure algometer, pressure will be applied to selected points until the patient experiences pain, at which point the test for that region will be terminated. The measurements will include bilateral thighs, the middle points of the pretibial region, and the control region (left forearm's volar surface). A Wagner manual pressure algometer (1 cm² probe - 10 kg/20 lb) will be used.

SECONDARY OUTCOMES:
Short Form-12 | 3 months
  The Short Form-12 is a short questionnaire used to assess individuals' physical and mental health. It is a shortened version of the Short form-36 and covers 8 health dimensions: physical function, social function, physical role limitations, emotional role limitations, mental health, general health, pain, and energy. The results are summarized into physical and mental health components, providing a quick and practical overview of general health status. A Turkish validity and reliability study has been conducted.
Lower Extremity Functional Scale, LEFS | 3 months
  The Lower Extremity Functional Scale (LEFS) is a tool used to assess the function of the lower extremities (legs, knees, hips, and feet). It measures the limitations in daily activities related to lower extremity function. It is used to monitor functional status after injury or illness, evaluate treatment response, and set treatment goals. The scale consists of 20 physical activities, rated from 0 (unable to perform) to 4 (no difficulty performing). A total score of 80 indicates a high functional level. A Turkish validity and reliability study has been conducted.
Bioelectrical Impedance Analysis | 3 months
  Bioelectrical Impedance Analysis is used to assess body composition, measuring parameters such as body fat percentage, muscle mass, water content, and metabolic age. It uses bioelectrical impedance analysis technology, sending a low-level electrical current through the body. Since different body components conduct this current in various ways, the resistance data obtained is used to determine fat, muscle, and water levels. Easy to use, these devices are typically in the form of a scale, and users can get results within seconds by stepping on the device. Widely preferred by athletes, dietitians, and individuals, these devices are considered reliable tools for monitoring health and achieving fitness goals.
Evaluation with ultrasonography | 3 months
  Subcutaneous fat thickness measurements for diagnosing lipedema are recommended at specific sites, including the mid-thigh, pretibial, lateral calf, and supramalleolar regions. Subcutaneous thickness, including the skin, is measured 6-8 cm above the medial malleolus. Even in cases of proximal lipedema, this measurement serves as a reliable reference. Based on these measurements: 12-15 mm indicates mild lipedema or lipohypertrophy, 15-20 mm indicates moderate lipedema, >20 mm indicates prominent lipedema, and >30 mm indicates severe lipedema.
Lower extremity measurements | 3 months
  For circumference calculation, measurements will be taken bilaterally at the mid-thigh, knee circumference, pretibial area, ankle, and proximal metatarsophalangeal joint.
  For volume calculation, measurements will be taken at 4 cm intervals starting from the ankle. The obtained circumference measurements will be converted into volume using an Excel worksheet.
Lower extremity volumetric measurements | 3 months
  Volume calculation with lower extremity circumference measurement at 4 cm intervals

CONTACTS AND LOCATIONS:
Overall Officials: Emre Ata, Assoc.Prof, Study Chair — Sultan Abdülhamid Han Research and Training Hospital
Locations (1):
- Sultan 2. Abdülhamid Han Eğitim ve Araştırma Hastanesi, İstanbul, Üsküdar 34000, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data sharing is not planned

REFERENCES:
- [Result] Chakraborty A, Crescenzi R, Usman TA, Reyna AJ, Garza ME, Al-Ghadban S, Herbst KL, Donahue PMC, Rutkowski JM. Indications of Peripheral Pain, Dermal Hypersensitivity, and Neurogenic Inflammation in Patients with Lipedema. Int J Mol Sci. 2022 Sep 7;23(18):10313. doi: 10.3390/ijms231810313. PMID 36142221
- [Result] Dinnendahl R, Tschimmel D, Low V, Cornely M, Hucho T. Non-obese lipedema patients show a distinctly altered quantitative sensory testing profile with high diagnostic potential. Pain Rep. 2024 Apr 11;9(3):e1155. doi: 10.1097/PR9.0000000000001155. eCollection 2024 Jun. PMID 38617100
- [Result] Soylu C, Kutuk B. Reliability and Validity of the Turkish Version of SF-12 Health Survey. Turk Psikiyatri Derg. 2022 Summer;33(2):108-117. doi: 10.5080/u25700. English, Turkish. PMID 35730511
- [Result] Jebb SA, Cole TJ, Doman D, Murgatroyd PR, Prentice AM. Evaluation of the novel Tanita body-fat analyser to measure body composition by comparison with a four-compartment model. Br J Nutr. 2000 Feb;83(2):115-22. doi: 10.1017/s0007114500000155. PMID 10743490
- [Result] Duzce Keles E, Birtane M, Ekuklu G, Kilincer C, Caliyurt O, Tastekin N, Is EE, Ketenci A, Neblett R. Validity and reliability of the Turkish version of the central sensitization inventory. Arch Rheumatol. 2021 Oct 18;36(4):518-526. doi: 10.46497/ArchRheumatol.2022.8665. eCollection 2021 Dec. PMID 35382371
- [Result] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Result] Amato ACM, Saucedo DZ, Santos KDS, Benitti DA. Ultrasound criteria for lipedema diagnosis. Phlebology. 2021 Sep;36(8):651-658. doi: 10.1177/02683555211002340. Epub 2021 Apr 15. PMID 33853452